CLINICAL TRIAL: NCT06763510
Title: Comparison of the Effects of Two Different Local Anesthetics Used in Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Ankara Ataturk Sanatorium Training and Research Hospital (Other Government)
Collaborators: Fatih University (Other)
Responsible Party: Principal Investigator, Azra Ozanbarci, specialist, Ankara Ataturk Sanatorium Training and Research Hospital
Other Study IDs: 26247029-514-04-01
Record Dates: First submitted 2024-12-31; First posted 2025-01-08 (Actual); Last update posted 2025-01-20 (Actual); Status verified 2025-01

CONDITIONS: Local Anaesthesia
Keywords: Spinal anesthesia; Local anesthetics; Thermoregulation; Baricity
MeSH Terms: interventions — Levobupivacaine; Bupivacaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Isobaric levobupivacaine
  Interventions: Drug: Chirocaine
- Hyperbaric bupivacaine
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: Chirocaine — Our study was conducted on forty full-term pregnant women scheduled for elective cesarean sections under spinal anesthesia. At an operating room temperature of twenty-four degrees Celsius, peripheral body temperature was measured using temperature probes attached to the lower medial parts of the same side's lower and upper extremities, and central body temperature was measured with a tympanic thermometer. Isobaric levobupivacaine was used in spinal anesthesia applications. After spinal anesthesia, tympanic temperature, arm and leg temperatures, mean arterial pressure, heart rate, and oxygen saturation were measured and recorded at baseline, the first, third, and fifth minutes, and every five minutes thereafter until the end of surgery.
  Other Names: levobupivacaine
  Groups: Isobaric levobupivacaine
Drug: Bupivacaine — Our study was conducted on forty full-term pregnant women scheduled for elective cesarean sections under spinal anesthesia. At an operating room temperature of twenty-four degrees Celsius, peripheral body temperature was measured using temperature probes attached to the lower medial parts of the same side's lower and upper extremities, and central body temperature was measured with a tympanic thermometer. Hyperbaric bupivacaine was used in spinal anesthesia applications. After spinal anesthesia, tympanic temperature, arm and leg temperatures, mean arterial pressure, heart rate, and oxygen saturation were measured and recorded at baseline, the first, third, and fifth minutes, and every five minutes thereafter until the end of surgery.
  Groups: Hyperbaric bupivacaine

SUMMARY:
Objective: This study aimed to compare the effects of two different local anesthetics with different baricity used in spinal anesthesia on thermoregulation.

Materials and Methods: The study was conducted on forty full-term pregnant women scheduled for elective cesarean sections under spinal anesthesia. At an operating room temperature of twenty-four degrees Celsius, peripheral body temperature was measured using temperature probes attached to the lower medial parts of the same side's lower and upper extremities, and central body temperature was measured with a tympanic thermometer. Isobaric levobupivacaine and hyperbaric bupivacaine were used in spinal anesthesia applications. After spinal anesthesia, tympanic temperature, arm and leg temperatures, mean arterial pressure, heart rate, and oxygen saturation were measured and recorded at baseline, the first, third, and fifth minutes, and every five minutes thereafter until the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Term pregnant with elective cesarean section planned under spinal anesthesia
* ASA I-II
* 18-40 years old

Exclusion Criteria:

* patients in whom spinal anesthesia is contraindicated,
* patients with neuromuscular disease,
* alcohol and substance abusers,
* patients with a body mass index (BMI) <18.5 kg/m² or >35 kg/m²,
* those taking medications that may affect thermoregulation such as vasodilators,
* patients with thyroid disease,
* patients with fever and infection,
* patients with known allergies to study drugs.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: The study was conducted on 40 full-term pregnant women aged 18-40, classified as ASA I-II, who were scheduled for elective cesarean sections under spinal anesthesia. All patients included in the study were informed and gave their written and verbal consent.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2015-02-01 (Actual); Primary Completion 2015-04-30 (Actual); Study Completion 2015-07-30 (Actual)

PRIMARY OUTCOMES:
Temperature | During operation
  Isobaric levobupivacaine or hyperbaric bupivacaine were used in spinal anesthesia applications. After spinal anesthesia, tympanic temperature, arm and leg temperatures were measured and recorded at the beginning, first, third and fifth minutes and then every five minutes until the end of the surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Fatih University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No